CLINICAL TRIAL: NCT05312671
Title: Atezolizumab With Platinum and Etoposide Chemotherapy Followed by Cystectomy for Patients With Localized Small Cell Neuroendocrine Bladder Cancer
Brief Title: Atezolizumab Plus Etoposide and Platinum in Small Cell Bladder Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: J2208; IRB00313218 (Other: JHM IRB); ML42154 (Other: Genentech)
Record Dates: First submitted 2022-03-28; First posted 2022-04-05 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Small Cell Neuroendocrine Carcinoma of Bladder; Bladder Cancer; Urothelial Carcinoma Bladder
Keywords: Small Cell Bladder Cancer; Atezolizumab; Cisplatin; Carboplatin; Platinum; Etoposide; Cystectomy
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — atezolizumab; Carboplatin; Cisplatin; Etoposide; Podophyllotoxin; Cystectomy

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Atezolizumab with Platinum and Etoposide, followed by cystectomy. (Experimental): The study population will include male and female patients over the age of 18 with invasive (cT1-cT4) small cell / neuroendocrine carcinoma of the bladder (MIBC), with or without urothelial cancer component, who are eligible for platinum based chemotherapy and immunotherapy. All patients will be fit to undergo surgical resection of their cancer by cystectomy. Patients with resectable N1 disease within the true pelvis are eligible.
  Atezolizumab will be administered by intravenous (IV) infusion at a fixed dose of 1200 mg Day 1 of every 21 day cycle with chemotherapy x 4 cycles. Following cystectomy, Atezolizumab maintenance Q 21 days will continue until unacceptable toxicity or loss of clinical benefit as determined by the investigator after an integrated assessment of radiographic and biochemical data, local biopsy results (if available), and clinical status (e.g., symptomatic deterioration such as pain secondary to disease), or up to 1 year (e.g., 16 cycles).
  Interventions: Drug: Atezolizumab; Drug: Carboplatin; Drug: Cisplatin; Drug: Etoposide; Procedure: Cystectomy

INTERVENTIONS:
Drug: Atezolizumab — Atezolizumab 20 mL (1200 mg) on Day 1, once every 3 weeks for up to 20 cycles (each cycle = 21 days)
  Other Names: Tecentriq
Drug: Carboplatin — Carboplatin AUC 5 IV on Day 1, once every 3 weeks for first 4 cycles (each cycle = 21 days).
  Other Names: CBDCA, Paraplatin, JM-8, NSC-241240
Drug: Cisplatin — Cisplatin 70 mg/m2 IV on Day 1, once every 3 weeks for first 4 cycles (each cycle = 21 days).
  Other Names: Cis-Diaminedichloroplatinum, CDDP
Drug: Etoposide — Etoposide 100 mg/m2 IV on Days 1 - 3 every cycle for the first 4 cycles (each cycle = 21 days)
  Other Names: VP-16, VePesid, VP-16-213, EPEG, epipodophyllotoxin, NSC # 141540
Procedure: Cystectomy — Cystectomy should be performed within 42 days after completion of last administered study therapy of induction phase (first 4 cycles of chemotherapy).

SUMMARY:
This is a single arm, Phase II trial involving the use of atezolizumab plus platinum and etoposide for patients with locally advanced urothelial cancer. The primary goal of this trial is to assess the pathologic complete response rate at cystectomy in patients after being treated with a combination therapy of atezolizumab, platinum, and etoposide.

DETAILED DESCRIPTION:
The study population will include male and female patients over the age of 18 with invasive (cT1-cT4) small cell / neuroendocrine carcinoma of the bladder (MIBC), with or without urothelial cancer component, who are eligible for platinum based chemotherapy and immunotherapy. All patients will be fit to undergo surgical resection of their cancer by cystectomy. Patients with resectable N1 disease within the true pelvis are eligible.

Participants will receive:

Atezolizumab 1,200 mg IV Day 1 Etoposide 100 mg/m2 IV on Days 1-3 Carboplatin AUC 5 IV on Day 1 or Cisplatin 70 mg/m2 IV on Day 1 (Patients can be switched at investigator's discretion between cisplatin and carboplatin between cycles. Rationale must be provided.) Repeat q 21 days x 4 cycles

Atezolizumab will be administered by intravenous (IV) infusion at a fixed dose of 1200 mg Day 1 of every 21 day cycle with chemotherapy x 4 cycles. Following cystectomy, Atezolizumab maintenance Q 21 days will continue until unacceptable toxicity or loss of clinical benefit as determined by the investigator after an integrated assessment of radiographic and biochemical data, local biopsy results (if available), and clinical status (e.g., symptomatic deterioration such as pain secondary to disease), or up to 1 year (e.g., 16 cycles).

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed invasive carcinoma of the bladder with pure, or any component of, small cell or high grade neuroendocrine features with or without urothelial cancer - localized ≥ cT1-T4aN1

A formalin-fixed paraffin-embedded (FFPE) tumor specimen in a paraffin block (preferred) or at least 15 slides containing unstained, freshly cut, serial sections should be submitted along with an associated pathology report prior to study enrollment. If less than 15 slides are available, the patient may still be eligible for the study, after Principal Investigator confirmation has been obtained.

If archival tumor tissue is unavailable or is determined to be unsuitable for required testing, tumor tissue must be obtained from a biopsy performed at screening.

* Medically fit to undergo chemotherapy, immunotherapy and cystectomy
* 18 years old at time of consent
* ECOG performance status of 0 or 1
* Adequate hematologic and end organ function, defined by the following laboratory results obtained within 14 days prior to randomization:
* ANC ≥ 1500 cells/μL without granulocyte colony-stimulating factor support
* Lymphocyte count ≥ 500/μL
* Platelet count ≥ 100,000/μL without transfusion
* Hemoglobin ≥ 9.0 g/dL -patients may be transfused to meet this criterion.
* INR or aPTT ≤ 1.5 × upper limit of normal (ULN) This applies only to patients who are not receiving therapeutic anticoagulation; patients receiving therapeutic anticoagulation should be on a stable dose.
* AST, ALT, and alkaline phosphatase ≤ 2.5 × ULN
* Serum bilirubin ≤ 1.5 × ULN Patients with known Gilbert disease who have serum bilirubin level ≤3 × ULN may be enrolled.
* Serum albumin >= 25 g/L (2.5 g/dL)
* Negative HIV test at screening (with the following exception: patients with a positive HIV test at screening are eligible provided they are stable on anti-retroviral therapy, have a CD4 count >= 200/µL, and have an undetectable viral load)
* Negative hepatitis B surface antigen (HBsAg) test at screening
* Negative total hepatitis B core antibody (HBcAb) test at screening, or positive total HBcAb test followed by a negative hepatitis B virus (HBV) DNA test at screening The HBV DNA test will be performed only for patients who have a negative HBsAg test and a positive total HBcAb test.
* Creatinine clearance >30. Patients receiving cisplatin must have creatinine clearance >50
* For women of childbearing potential (WOCBP): agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive methods, and agreement to refrain from donating eggs, as defined below:
* Women must remain abstinent or use contraceptive methods with a failure rate of <1% per year during the treatment period and for 5 months after the final dose of atezolizumab and for 30 days after the final dose of cisplatin/ carboplatin and etoposide. Women must refrain from donating eggs during this same period.
* A woman is considered to be of childbearing potential if she is postmenarchal, has not reached a postmenopausal state (>= 12 continuous months of amenorrhea with no identified cause other than menopause), and has not undergone surgical sterilization (removal of ovaries and/or uterus). The definition of childbearing potential may be adapted for alignment with local guidelines or requirements.
* Examples of contraceptive methods with a failure rate of < 1% per year include bilateral tubal ligation, male sterilization, hormonal contraceptives that inhibit ovulation, hormone-releasing intrauterine devices, and copper intrauterine devices.

The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or postovulation methods) and withdrawal are not adequate methods of contraception.

* For men: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive measures, and agreement to refrain from donating sperm, as defined below:
* With a female partner of childbearing potential who is not pregnant, or a pregnant female partner men who are not surgically sterile must remain abstinent or use a condom plus an additional contraceptive method that together result in a failure rate of < 1% per year during the treatment period and for 8 months after the final dose of atezolizumab and 120 days after the final dose of etoposide. Men must refrain from donating sperm during this same period.
* The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or postovulation methods) and withdrawal are not adequate methods of contraception.
* Patients who give a written informed consent obtained according to local guidelines
* Patients who received mineralocorticoids (e.g., fludrocortisone), corticosteroids for chronic obstructive pulmonary disease (COPD) or asthma, or low-dose corticosteroids for orthostatic hypotension or adrenal insufficiency are eligible for the study.

Exclusion Criteria:

* No prior systemic treatment for small-cell bladder cancer (SCBC)
* Patients with concurrent upper urinary tract (i.e. ureter, renal pelvis) invasive urothelial carcinoma. (NOTE: Patients with history of non-invasive (Ta, Tis) upper tract urothelial carcinoma that has been definitively treated with at least one post- treatment disease assessment (i.e. cytology, biopsy, imaging) that demonstrates no evidence of residual disease are eligible). Individual cases will be discussed at investigator discretion.
* Patients with another active second malignancy other than non-melanoma skin cancers and biochemical relapsed prostate cancer. Patients that have completed all necessary therapy and are considered to be at less than 30% risk of relapse are not considered to have an active second malignancy and are eligible for enrollment.
* Patients who have received prior systemic chemotherapy for urothelial bladder cancer.

Prior BCG and intravesical chemotherapy are allowed

* Any metastatic disease including leptomeningeal disease or brain metastasis on baseline brain imaging
* Uncontrolled tumor-related pain - Patients requiring pain medication must be on a stable regimen at study entry.

Patients requiring pain medication must be on a stable regimen at study entry.

Uncontrolled or symptomatic hypercalcemia (ionized calcium > 1.5 mmol/L, calcium > 12 mg/dL or corrected serum calcium > ULN

* Active or history of autoimmune disease or immune deficiency, including, but not limited to, myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, antiphospholipid antibody syndrome, Wegener granulomatosis, Sjögren syndrome, Guillain-Barré syndrome, or multiple sclerosis, with the following exceptions:
* Patients with a history of autoimmune-related hypothyroidism who are on thyroid- replacement hormone are eligible for the study.
* Patients with controlled Type 1 diabetes mellitus who are on an insulin regimen are eligible for the study.
* Patients with eczema, psoriasis, lichen simplex chronicus, or vitiligo with dermatologic manifestations only (e.g., patients with psoriatic arthritis are excluded) are eligible for the study provided all of following conditions are met:
* Rash must cover < 10% of body surface area
* Disease is well controlled at baseline and requires only low-potency topical corticosteroids
* No occurrence of acute exacerbations of the underlying condition requiring psoralen plus ultraviolet A radiation, methotrexate, retinoids, biologic agents, oral calcineurin inhibitors, or high-potency or oral corticosteroids within the previous 12 months
* Individual cases can be discussed at investigator discretion. Refer to Appendix H for more details
* History of idiopathic pulmonary fibrosis, organizing pneumonia (e.g., bronchiolitis obliterans), drug-induced pneumonitis, or idiopathic pneumonitis, or evidence of active pneumonitis on screening chest computed tomography (CT) scan. History of radiation pneumonitis in the radiation field (fibrosis) is permitted.
* Active tuberculosis
* Significant cardiovascular disease (such as New York Heart Association Class II or greater cardiac disease, myocardial infarction, or cerebrovascular accident) within 3 months prior to initiation of study treatment, unstable arrhythmia, or unstable angina
* Patients who have undergone major surgery (e.g. intra-thoracic, intra- abdominal or intra-pelvic), open biopsy or significant traumatic injury ≤ 4 weeks prior to starting study drug, or patients who have had minor procedures (i.e. TURBT), percutaneous biopsies or placement of vascular access device ≤1 week prior to starting study drug, or who have not recovered from side effects of such procedure or injury
* History of malignancy other than small cell bladder cancer within 5 years prior to screening, with the exception of malignancies with a negligible risk of metastasis or death (e.g., 5-year OS rate > 90%), such as adequately treated carcinoma in situ of the cervix, non melanoma skin carcinoma, localized prostate cancer, ductal carcinoma in situ, or Stage I uterine cancer
* Severe infection within 4 weeks prior to initiation of study treatment, including, but not limited to, hospitalization for complications of infection, bacteremia, or severe pneumonia
* Treatment with therapeutic oral or IV antibiotics within 2 weeks prior to initiation of study treatment. Patients receiving prophylactic antibiotics (e.g., to prevent a urinary tract infection or chronic obstructive pulmonary disease exacerbation) are eligible for the study.
* Prior allogeneic stem cell or solid organ transplantation
* Any other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding that contraindicates the use of an investigational drug, may affect the interpretation of the results, or may render the patient at high risk from treatment complications
* Treatment with a live, attenuated vaccine (e.g., FluMist®) within 4 weeks prior to initiation of study treatment, or anticipation of need for such a vaccine during atezolizumab treatment or within 5 months after the final dose of Atezolizumab
* Current treatment with anti-viral therapy for HBV
* Treatment with investigational therapy within 28 days prior to initiation of study treatment
* Prior treatment with CD137 agonists or other immune checkpoint blockade therapies, including anti-CTLA-4, anti-PD-1, and anti-PD-L1 therapeutic antibodies
* Treatment with systemic immunostimulatory agents (including, but not limited to, interferon and interleukin 2 [IL-2]) within 4 weeks or 5 half-lives of the drug (whichever is longer) prior to initiation of study treatment
* Treatment with systemic immunosuppressive medication (including, but not limited to, corticosteroids, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti- TNF-α agents) within 2 weeks prior to initiation of study treatment, or anticipation of need for systemic immunosuppressive medication during study treatment.
* Patients who received acute, low-dose systemic immunosuppressant medication or a one-time pulse dose of systemic immunosuppressant medication (e.g., 48 hours of corticosteroids for a contrast allergy) are eligible for the study after Principal Investigator confirmation has been obtained.
* History of severe allergic anaphylactic reactions to chimeric or humanized antibodies or fusion proteins
* Known hypersensitivity to Chinese hamster ovary cell products or to any component of the atezolizumab formulation
* Known allergy or hypersensitivity to any component of Cisplatin, carboplatin or etoposide
* Pregnancy or breastfeeding, or intention of becoming pregnant during study treatment or within 5 months of atezolizumab after the final dose of study treatment. Women of childbearing potential must have a negative serum pregnancy test result within 14 days prior to initiation of study treatment.
* Patients who have had radiotherapy to the bladder, or radiotherapy ≤ 4 weeks prior to starting study drug, or who have not recovered from radiotherapy toxicities

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Estimated)
Dates: Start 2022-06-27 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2029-10 (Estimated)

PRIMARY OUTCOMES:
Pathologic complete response (ypCR) at cystectomy | up to 18 months
  The number of participants with pathological complete responses (ypCR) at cystectomy. Pathologic complete response is defined as post-treatment cystectomy tumor stages N0 and M0, with T-stage T0.

SECONDARY OUTCOMES:
Number of participants with non-muscle invasive disease | up to 18 months
  Non-muscle invasive disease is defined as <ypT1N0 at cystectomy.
Safety and tolerability of combination chemotherapy and cystectomy as assessed by number of participants experiencing adverse events | 4.5 years
  Number of participants experiencing dose limiting toxicities and treatment-related adverse events, as defined by Common Terminology Criteria for Adverse Events Version 5.0 (CTCAE v5.0).
Incidence of brain metastases in follow-up | up to 5 years
  Number of participants who develop brain metastases during follow-up
1-year overall survival rate (1-yr OS) | up to 4 years
  Number of participants alive 1 year after last dose
2-year overall survival rate (2-yr OS) | up to 5 years
  Number of participants alive 2 years after last dose
Disease Free Survival | up to 5 years
  Number of participants without disease recurrence
Feasibility of atezolizumab administration with platinum and etoposide chemotherapy prior to surgery | up to 18 months
  Number of participants during the first stage of the study (first 15 patients) proceeding to surgery without extended treatment related delays.

CONTACTS AND LOCATIONS:
Overall Officials: Jean Hoffman-Censits, MD, Principal Investigator — Johns Hopkins University
Locations (2):
- United States (2):
  - Johns Hopkins University: Sibley Memorial Hospital, Washington D.C., District of Columbia
  - Johns Hopkins University: Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland

IPD SHARING:
Plan to Share IPD: No